CLINICAL TRIAL: NCT07013955
Title: Comparative Study Between the Effect of Nasal Packing With Dexmedetomidine, Midazolam or Bupivacaine on Surgical Field Visualization During Functional Endoscopic Sinus Surgery .
Brief Title: Comparative Study Between the Effect of Dexmedetomidine ,Midazolam or Bupivacaine Packing During FESS on Surgical Field Visualization
Acronym: FESS (Function
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Fatma Rabea Mohammed, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1465/02/2025
Record Dates: First submitted 2025-05-16; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-02

CONDITIONS: Surgical Hemostasis
MeSH Terms: interventions — Sodium Chloride; Dexmedetomidine; Midazolam; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Group I (Group C): (control group) Patients in this group will receive only 5 ml of intranasal saline.
  Group II (Group D): Patients in this group will receive only intranasal Dexmedetomidine (1 mcg/kg) made up to 5 ml in normal saline.
  Group III (Group M): Patients in this group will receive only intranasal midazolam (0.2 mg/kg) made up to 5 ml in normal saline.
  Group IV (Group B): Patients in this group will receive only intranasal bupivacaine (0.5% solution) 5 ml.
Who Masked: Participant, Care Provider
Masking Description: Group I (Group C): (control group) Patients in this group will receive only 5 ml of intranasal saline.
  Group II (Group D): Patients in this group will receive only intranasal Dexmedetomidine (1 mcg/kg) made up to 5 ml in normal saline.
  Group III (Group M): Patients in this group will receive only intranasal midazolam (0.2 mg/kg) made up to 5 ml in normal saline.
  Group IV (Group B): Patients in this group will receive only intranasal bupivacaine (0.5% solution) 5 ml.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group I (Group C): (control group) (Placebo Comparator): Patients in this group will receive only 5 ml of intranasal saline.
  Interventions: Drug: Saline
- Group II (Group D) (Active Comparator): Patients in this group will receive only intranasal Dexmedetomidine (1 mcg/kg) made up to 5 ml in normal saline.
  Interventions: Drug: Dexmedetomidine
- Group III (Group M) (Active Comparator): Patients in this group will receive only intranasal midazolam (0.2 mg/kg) made up to 5 ml in normal saline.
  Interventions: Drug: Midazolam
- Group IV (Group B) (Active Comparator): Patients in this group will receive only intranasal bupivacaine (0.5% solution) 5 ml.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Saline — Group I (Group C): (control group) Patients in this group will receive only 5 ml of intranasal saline.
  Arms: Group I (Group C): (control group)
Drug: Dexmedetomidine — Group II (Group D): Patients in this group will receive only intranasal Dexmedetomidine (1 mcg/kg) made up to 5 ml in normal saline.
  Arms: Group II (Group D)
Drug: Midazolam — Group III (Group M): Patients in this group will receive only intranasal midazolam (0.2 mg/kg) made up to 5 ml in normal saline.
  Arms: Group III (Group M)
Drug: Bupivacaine — Group IV (Group B): Patients in this group will receive only intranasal bupivacaine (0.5% solution) 5 ml.
  Arms: Group IV (Group B)

SUMMARY:
The goal of this interventional study is to compare the nasal packing with dexmedetomidine .midazolam or bupivacaine on surgical field visualization during FESS . Study groups :

Group I (Group C): (control group) Patients in this group will receive only 5 ml of intranasal saline.

Group II (Group D): Patients in this group will receive only intranasal Dexmedetomidine (1 mcg/kg) made up to 5 ml in normal saline.

Group III (Group M): Patients in this group will receive only intranasal midazolam (0.2 mg/kg) made up to 5 ml in normal saline.

Group IV (Group B): Patients in this group will receive only intranasal bupivacaine (0.5% solution) 5 ml.

DETAILED DESCRIPTION:
This study will be conducted in Minia University Hospital This prospective randomized double-blind controlled clinical study will be conducted on 144 adult patients of both sexes, aged between 16 and 60 years old, with BMI up to 30 with ASA physical status I & II.

Parameters assessed:

* Intraoperative Monitoring:

  1. Surgical field visualization using the Boezaart scale.
  2. Hemodynamic changes among the study groups including the heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MAP), and oxygen saturation (SPO2) measured at baseline, (10 min after packing), every 5 mins till the end of the surgery.
* Postoperative Evaluation

  1. Assess postoperative pain using VAS every 1 hour for the 1st six hours, every 2 hours for 12 hours then every 4 hours till 24 hours postoperatively.
  2. The sedation score will be assessed using the Ramsay sedation score as VAS intervals.
  3. Surgeon satisfaction will be assessed by a Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* aged between 16 and 60 years old
* with BMI up to 30
* with ASA physical status I & II.

Exclusion Criteria:

* Patients with a history of allergy to the study drugs.
* Pregnant and lactating females.
* Patients with severe liver, renal, or cardiac diseases
* Patients with repeated nasal surgeries.
* Patients with psychiatric conditions.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
We aim to assess the efficacy of intranasal packing with dexmedetomidine, midazolam, or bupivacaine in reducing bleeding during FESS operations in patients who require general anesthesia with endotracheal intubation. | Intraoperative (for 2 hours maximally)
  Evaluate the efficacy of intranasal packing with dexmedetomidine, midazolam, or bupivacaine in improving surgical field visualization using the Boezaart Score.
  Grade Assessment 0 No bleeding (cadaveric conditions)
  1. Slight bleeding, no suctioning required
  2. Slight bleeding, occasional suctioning required
  3. Slight bleeding, frequent suctioning required; bleeding threatens the surgical field a few seconds after suction is removed
  4. Moderate bleeding, frequent suctioning required, and bleeding threatens the surgical field directly after suction is removed
  5. Severe bleeding, constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely threatened and surgery usually not possible

SECONDARY OUTCOMES:
Total requirement of nitroglycerine as a hypotensive agent. | postoperative (at the end of operation after 2 hours )
  Intraoperative total requirement of nitroglycerine as a hypotensive agent.
Comparing the surgeon satisfaction among the study groups. | Postoperative (immediately at the end of the surgery )
  Surgeon satisfaction will be assessed by a Likert scale Score 1 (very poor) Uncontrollable bleeding Score 2 (poor) Severe bleeding requiring repeated suctioning, with the quality of the field collapsing immediately after suctioning Score 3 (satisfactory) Moderate bleeding requiring intermittent suctioning. Score 4 (good) Partial bleeding, sometimes requiring suctioning the quality of the surgical field was good.
  Score 5 (excellent) No bleeding/bloodless field; the surgery field was excellent
Hemodynamic changes among the study groups: | Intraoperative (baseline then every 5 minutes till the end of surgery )
  2.Hemodynamic changes among the study groups including the heart rate (HR) in beat per minute, systolic blood pressure (SBP) in mmHg, diastolic blood pressure (DBP) in mmHg, mean blood pressure (MAP) in mmHg, and oxygen saturation (SPO2) in percentage measured at baseline, (10 min after packing), every 5 mins till the end of the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma R Mohammed, MD, Principal Investigator — Minia University
Locations (1):
- Faculty of Medicine, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No
Data is available with corresponding authors on reasonable request